CLINICAL TRIAL: NCT03627910
Title: Pressure Ulcers in Patients Receiving Enteral Nutrition Therapy. What is the Relationship With Gut Microbiota?
Brief Title: Pressure Ulcers in Patients Receiving Enteral Nutrition Therapy and Their Relationship With Gut Microbiota
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ulcere1_FDG
Record Dates: First submitted 2018-08-01; First posted 2018-08-14 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Malnutrition; Pressure Ulcer
Keywords: gut microbiota; Iatrogenic malnutrition; pressure ulcer
MeSH Terms: conditions — Malnutrition; Pressure Ulcer | interventions — Zinc; Arginine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Participants assigned to the treatment group will be administered a commercial symbiotic (Probinul Ca.Di.GROUP S.r.l.) for the entire duration of the study (90 days) plus an enteral nutrition formula rich in zinc and arginine
  Interventions: Dietary Supplement: symbiotic; Dietary Supplement: zinc and arginine
- Control group (Active Comparator): Control group will be administered only an enteral nutrition formula rich in zinc and arginine
  Interventions: Dietary Supplement: zinc and arginine

INTERVENTIONS:
Dietary Supplement: symbiotic — Feed supplementation
  Arms: Treatment group
Dietary Supplement: zinc and arginine — Feed supplementation

SUMMARY:
Participants will be randomly assigned to the experimental group where they will be given enteral nutrition formula rich in zinc and arginine plus a symbiotic (Probinul- Ca.Di.GROUP S.r.l.) once a day for 90 days or the control group where they will receive only the enteral nutrition formula rich in zinc and arginine.

DETAILED DESCRIPTION:
Participants belonging to both experimental and control group will be evaluated at admission (T0), 45 days after admission (T45) and at the end of the study (T90, 90 days after admission). At each time point patients' nutritional status will be determined and the following biochemical parameters will be investigated: lymphocyte count, total proteins, protidogram, prealbumin, transferrin, vascular endothelial growth factor (VEGF), Platelet-derived growth factor (PDGF), beta transforming growth factor (TGF-beta). Analysis of fecal DNA will be also performed to characterize the gut microbiota. In addition, at the baseline and at T45 participants will be administered the Braden scale for predicting pressure sore risk.

ELIGIBILITY:
Inclusion Criteria:

* Patients with enteral nutrition therapy
* Presence of pressure ulcers
* Previous antibiotic therapy

Exclusion Criteria:

* nutrition per os
* absence of pressure ulcers
* absence of previous antibiotic therapy

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-06-11 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Determination of Transforming Growth Factor β (TGF-β1), Epidermal Growth Factor (EGF) and Vascular Endothelial Growth Factor (VEGF) | 90 days after the fist time point (baseline assessment)
  Human EGF, human VEGF/human TGF-β1 will be measured on aliquots (20 μl) of plasma using Quantikine® ELISA Human Immunoassay (R&D System, Abingdon, UK), following the manufacturer's protocol. The quantitative sandwich enzyme immunoassay technique will be used. A monoclonal antibody specific for human EGF/human VEGF, is pre-coated onto a microplate. For TGF -β1 assay latent TGF-β1 must be activated before test, following a procedure of acidification and then neutralization to pH 7.2-7.6. Standards and samples are pipetted into the wells and EGF or VEGF present is bound by the immobilized antibody. After washing away unbound substances, an enzyme-linked polyclonal antibody specific for human EGF/human VEGF is added to the wells. After removing any unbound antibody-enzyme reagent, a substrate solution is added and colour develops in proportion to the amount of EGF bound. Colour development is stopped, and colour intensity measured. Tests will be performed in triplicates for each sample.

SECONDARY OUTCOMES:
Monitoring modification of gut microbiota through DNA extraction and quantification | 45 days after the fist time point (baseline assessment) and 90 days after the fist time point (baseline assessment)
  Total DNA will be extracted in triplicate from all the fecal samples by following the QIAamp DNA Stool Mini Kit instructions (Qiagen) and quantified with a Qubit® 2.0 fluorometer (Invitrogen, USA). Molecular weight and fragment length of DNA will be checked on 1.5 % agarose gel; the yield will be calculated as µg DNA/g feces. Quantitative PCR (qPCR) assays will be conducted using the specific primers rpoB1, rpoB1o and rpoB2 that generate amplicons of 250-bp, on 10 ng DNA templates for all the samples. Amplification will be carried out and three simultaneous replicates will be carried out for each of analyzed sample.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luisa Eliana Luisi, MD, Study Chair — Don Gnocchi Foundation, Italy
Locations (1):
- Fondazione Don Carlo Gnocchi, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fan Y, Pedersen O. Gut microbiota in human metabolic health and disease. Nat Rev Microbiol. 2021 Jan;19(1):55-71. doi: 10.1038/s41579-020-0433-9. Epub 2020 Sep 4. PMID 32887946
- [Background] Munoz N, Posthauer ME, Cereda E, Schols JMGA, Haesler E. The Role of Nutrition for Pressure Injury Prevention and Healing: The 2019 International Clinical Practice Guideline Recommendations. Adv Skin Wound Care. 2020 Mar;33(3):123-136. doi: 10.1097/01.ASW.0000653144.90739.ad. PMID 32058438
- [Background] Luisi MLE, Lucarini L, Biffi B, Rafanelli E, Pietramellara G, Durante M, Vidali S, Provensi G, Madiai S, Gheri CF, Masini E, Ceccherini MT. Effect of Mediterranean Diet Enriched in High Quality Extra Virgin Olive Oil on Oxidative Stress, Inflammation and Gut Microbiota in Obese and Normal Weight Adult Subjects. Front Pharmacol. 2019 Nov 15;10:1366. doi: 10.3389/fphar.2019.01366. eCollection 2019. PMID 31803056
- [Background] Cereda E, Neyens JCL, Caccialanza R, Rondanelli M, Schols JMGA. Efficacy of a Disease-Specific Nutritional Support for Pressure Ulcer Healing: A Systematic Review and Meta-Analysis. J Nutr Health Aging. 2017;21(6):655-661. doi: 10.1007/s12603-016-0822-y. PMID 28537329
- [Background] Lynch SV, Pedersen O. The Human Intestinal Microbiome in Health and Disease. N Engl J Med. 2016 Dec 15;375(24):2369-2379. doi: 10.1056/NEJMra1600266. No abstract available. PMID 27974040
- [Background] Valentini L, Pinto A, Bourdel-Marchasson I, Ostan R, Brigidi P, Turroni S, Hrelia S, Hrelia P, Bereswill S, Fischer A, Leoncini E, Malaguti M, Blanc-Bisson C, Durrieu J, Spazzafumo L, Buccolini F, Pryen F, Donini LM, Franceschi C, Lochs H. Impact of personalized diet and probiotic supplementation on inflammation, nutritional parameters and intestinal microbiota - The "RISTOMED project": Randomized controlled trial in healthy older people. Clin Nutr. 2015 Aug;34(4):593-602. doi: 10.1016/j.clnu.2014.09.023. Epub 2014 Oct 8. PMID 25453395
- [Background] Ammons MC, Morrissey K, Tripet BP, Van Leuven JT, Han A, Lazarus GS, Zenilman JM, Stewart PS, James GA, Copie V. Biochemical association of metabolic profile and microbiome in chronic pressure ulcer wounds. PLoS One. 2015 May 15;10(5):e0126735. doi: 10.1371/journal.pone.0126735. eCollection 2015. PMID 25978400
- [Background] Wang X, Dong Y, Han X, Qi XQ, Huang CG, Hou LJ. Nutritional support for patients sustaining traumatic brain injury: a systematic review and meta-analysis of prospective studies. PLoS One. 2013;8(3):e58838. doi: 10.1371/journal.pone.0058838. Epub 2013 Mar 19. PMID 23527035
- [Background] Teno JM, Gozalo P, Mitchell SL, Kuo S, Fulton AT, Mor V. Feeding tubes and the prevention or healing of pressure ulcers. Arch Intern Med. 2012 May 14;172(9):697-701. doi: 10.1001/archinternmed.2012.1200. PMID 22782196
- [Background] Ohura T, Nakajo T, Okada S, Omura K, Adachi K. Evaluation of effects of nutrition intervention on healing of pressure ulcers and nutritional states (randomized controlled trial). Wound Repair Regen. 2011 May-Jun;19(3):330-6. doi: 10.1111/j.1524-475X.2011.00691.x. PMID 21539650